CLINICAL TRIAL: NCT00713440
Title: Incretin Physiology and Beta-Cell Function Before and After Treatment With Steroid Hormone in Healthy Individuals
Brief Title: Incretin Physiology Associated With Steroid Hormone Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Katrine Bagge Hansen, MD, Glostrup University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ST-INK
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Type 2 Diabetes Mellitus; Steroids
Keywords: Incretin Effect; Steroids; Glucagon-Like Peptide 1; Gastric Inhibitory Peptide; Glucose-dependent Insulinotropic Polypeptide; Insulin; C-peptide; Glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Glucose Tolerance Test; Prednisolone; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 10 healthy Caucasian subjects without family history of diabetes
  Interventions: Other: Oral glucose test (OGTT); isoglycaemic iv. clamp; liquid meal test; Gastric Emptying Rate; Prednisolone; Paracetamol

INTERVENTIONS:
Other: Oral glucose test (OGTT); isoglycaemic iv. clamp; liquid meal test; Gastric Emptying Rate; Prednisolone; Paracetamol — OGTT: The test is performed with 50 g of glucose deluded in 300 ml. of water. Isoglycaemic iv. clamp: Iv glucose infusion mimicking the glucose response curve of the OGTT.
  Liquid Meal Test: The test is performed with 100g of formula milk in 300 ml. of water.
  Gastric Emptying Rate: Paracetamol absorption test. Adrenocortical Steroids: Use of 37,5 mg./day of prednisolone during 10 days
  Other Names: Prednisolone; Paracetamol

SUMMARY:
The purpose of this study is to evaluate whether the reduced incretin effect and the paradoxical glucagon responses during oral glucose ingestion and isoglycaemic iv glucose infusion observed in patients with type 2 diabetes are causes (non-inducible in lean healthy subjects without family history of diabetes) or consequences (inducible) of the diabetic state.

DETAILED DESCRIPTION:
The incretin effect is severely reduced in patients with type 2 diabetes. This pathophysiological trait is accompanied by an almost abolished insulinotropic effect of the incretin hormone glucose-dependent insulinotropic polypeptide (GIP) and a reduced insulinotropic potency of the other incretin hormone glucagon-like peptide-1 (GLP-1). Furthermore, recent studies suggest that hypersecretion of glucagon during oral glucose ingestion, as opposed to a normal suppression of glucagon during isoglycaemic intravenous (iv) administered glucose, further attenuates the incretin effect in patients with type 2 diabetes.

However, it remains unclear whether the severely reduced incretin effect and its accompanying pathophysiological traits characterizing patients with type 2 diabetes can be induced temporarily in healthy subjects by a short period of glucose homeostatic dysregulation.

In this study the incretin effect will be measured using 50-g oral glucose tolerance test and isoglycaemic iv glucose infusion and meal test in 10 healthy Caucasian subjects without family history of diabetes before and after dysregulation of glucose homeostasis using high calorie diet, physical inactivity and administration of adrenocortical steroids

ELIGIBILITY:
Inclusion Criteria:

* Caucasians without Type 2 or Type 1 Diabetes
* Normal OGTT (75 g of glucose) according to WHO criteria
* Normal hemoglobin
* Normal blood pressure

Exclusion Criteria:

* Liver disease
* Kidney disease
* Relatives (parents/siblings) with type 2 diabetes
* Pregnancy
* Contra-indications to treatment with adrenocortical steroids

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Incretin effect before and after dysregulation of glucose homeostasis using high calorie diet, physical inactivity and administration of adrenocortical steroids. | One year

SECONDARY OUTCOMES:
GLP-1 and GIP response curves | One year

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD; Ph-D, Study Director — Gentofte University Hospital; Tina Vilsboll, MD; Ph-D, DMSc, Study Chair — University of Copenhagen; Katrine B Hansen, MD, Principal Investigator — Glostrup University Hospital; Steen Larsen, MD; DMSc, Study Chair — Glostrup University Hospital; Jens J Holst, Professor: DMSc, Study Chair — University of Copenhagen
Locations (1):
- Clinical Physiology Department; Glostrup Univesity Hospital, Glostrup Municipality, Capital Region, Denmark

REFERENCES:
- [Derived] Hansen KB, Vilsboll T, Bagger JI, Holst JJ, Knop FK. Increased postprandial GIP and glucagon responses, but unaltered GLP-1 response after intervention with steroid hormone, relative physical inactivity, and high-calorie diet in healthy subjects. J Clin Endocrinol Metab. 2011 Feb;96(2):447-53. doi: 10.1210/jc.2010-1605. Epub 2010 Nov 3. PMID 21047927